CLINICAL TRIAL: NCT04656847
Title: Assessment of the Efficacy, Adherence and Tolerability of the Single Pill Combination Bisoprolol/PerindopRil In Patients With Previous Myocardial Infraction With Arterial Hypertension in the Daily Clinical practicE
Brief Title: PRIDE. Assessment of the Efficacy, Adherence and Tolerability of the Single Pill Combination Bisoprolol/Perindopril
Acronym: PRIDE
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05150-065-RUS
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Arterial Hypertension
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: in daily everyday routine practice — patients with HTN and CAD treated with the the single pill combination bisoprolol/perindopril for 12 weeks in the daily clinical practice Retrospective screening and evaluation of patient's eligibility to inclusion/ exclusion criteria for entering the study allows mitigating a potential risk of deliberative medicine administration within the observational program.
  Other Names: Baseline data will be collected retrospectively from medical records of stable CAD patients with HTN and a history of MI, including disease history of the patient.

SUMMARY:
This non-interventional, ambispective study was aimed at evaluating the effectiveness, safety, and tolerability of bisoprolol and perindopril SPC in previous myocardial infarction patients with HTN and CAD treated with the drug for 12 weeks in the daily clinical practice. SPC will be used according to the approved instruction for medical use of the medicine.

This is a multi-centre, observational, incomparative, ambispective study, which will retrospectively and prospectively collect clinical variables and socio-demographic data from medical records of patients with HTN and previous MI initiated with bisoprolol/perindopril SPC in real life settings.

DETAILED DESCRIPTION:
This is a multi-centre, observational, incomparative, ambispective study, which will retrospectively and prospectively collect clinical variables and socio-demographic data from medical records of patients with HTN and previous MI initiated with bisoprolol/perindopril SPC in real life settings.

Baseline data will be collected retrospectively from medical records of stable CAD patients with HTN and a history of MI, including disease history of the patient. To be included in the study for further prospective observation a patient should have been administered bisoprolol/ perindopril SPC within first three months before the Index Date. (Fig.1). Therefore, criteria for non-inclusion or inclusion of the patient in the study are to be retrospectively evaluated by the investigator using recorded clinical data available from medical records. Once a physician makes decision to include a patient in the study and, in particular, on the prospective observation for 3 months, a visit to the clinic for obtaining signed patient's consent to participate in the study should be appointed and made within 1 month from the Index Date.

Retrospective screening and evaluation of patient's eligibility to inclusion/ exclusion criteria for entering the study allows mitigating a potential risk of deliberative medicine administration within the observational program. Such studies are carried out in case of observational programs when the studied drug is administered in line with indications according to the instruction for its medical use.

Several multicenter, non-interventional, open, incomparable studies have been performed with bisoprolol/perindopril SPC in patients with HTN and coronary heart disease. A total of 70 general practitioners and cardiologists from primary care facilities will participate in the program. Each doctor will include about 7-8 patients. In total, it is planned to include at least 500 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina pectoris of class I-III according to the Canadian Cardiovascular Society (CCS) classification and a history of myocardial infarction no earlier (not less) than 3 months before inclusion in the study.

HTN (including resistant* hypertension)

* Signed informed consent to participate in the study.
* Bisoprolol/ perindopril SPC prescription** within 3 month period before Index date

Exclusion Criteria:

* Hypersensitivity to bisoprolol, perindopril, excipients of the medicine, or other ACE inhibitors.
* Any contraindication for bisoprolol/perindopril's SPC according to the instruction for medical use
* CAD, angina pectoris of functional class IV according to the CCS classification (Appendix 1).
* Chronic heart failure of class III-IV according to the New York Heart Association (NYHA) functional classification of heart failure (Appendix 3).
* Cerebrovascular diseases (ischemic, haemorrhagic stroke, or transient ischemic attack) within the past 6 months prior to inclusion in the study.
* A history of revascularization procedure within 3 months prior to inclusion in the study.
* Hypertrophic obstructive cardiomyopathy.
* Office BP ≥ 180/110 mm Hg on treatment
* Type 1 diabetes mellitus and decompensated type 2 diabetes mellitus.
* Bradycardia with a heart rate of less than 60 beats per minute.
* Atrioventricular block (II-III degree), sinoatrial block, or sick sinus syndrome.
* Severe bronchial asthma or severe chronic obstructive pulmonary disease.
* Arterial hypotension (BP less than 100/70 mm Hg).
* Pregnancy, breastfeeding.
* Secondary hypertension.
* Severe decompensated diseases of organs and systems requiring continuous treatment.
* Current participation in another clinical trial and within 30 days prior to signing informed consent.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: CAD patients with previous MI and HTN
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhanna Kobalava, Professor, Principal Investigator
Locations (1):
- Peoples' Friendship University of Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kobalava Z, Kvasnikov B, Burtsev Y; PRIDE study investigators. Effectiveness and Tolerability of Bisoprolol/Perindopril Single-Pill Combination in Patients with Arterial Hypertension and a History of Myocardial Infarction: The PRIDE Observational Study. Adv Ther. 2023 Jun;40(6):2725-2740. doi: 10.1007/s12325-023-02462-9. Epub 2023 Apr 8. PMID 37029871

RESULTS

PARTICIPANT FLOW:
Groups:
- CAD Patients With Previous MI and HTN: Observational study - 1 group - bisoprolol/perindopril FDC: single-pill combination of beta-blocker and ACE inhibitor
Period: 1 Month After Inclusion
Arm/Group | CAD Patients With Previous MI and HTN
Started | 504
Lipid Lowering Therapy | 463
Completed | 504
Not Completed | 0
Period: 3 Month After Inclusion
Arm/Group | CAD Patients With Previous MI and HTN
Started | 504
3 Month After Inclusion | 504
Lipid Lowering Therapy (Proportion of patients who were taking lipid lowering therapy (LLT) at week 12 of treatment) | 463
Completed (The study enrolled 504 patients. Of them, 481 (95.44%) were included in the population for full analysis set (FAS ).) | 481
Not Completed | 23
Not completed — lack of data on myocardial infarction and/or data by visits | 23

BASELINE CHARACTERISTICS:
Population: The study enrolled 504 patients. Of them, 481 (95.44%) were included in the population for analysis. Withdrawal of 23 patients occurred due to lack of data on myocardial infarction and/or data by visits of the study.
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.38 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 327
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 481

OUTCOME MEASURES:

1. Primary Outcome: Antihypertensive Effectiveness (SBP and DBP) of Bisoprolol/Perindopril SPC in CAD Patients With Previous MI and HTN at Week 12 of Treatment Compared With Baseline
Description: Change in the mean systolic and diastolic BP levels at week 12 of treatment with SPC compared with baseline among patients included in the study.
Time Frame: 3 months
Population: Changes in the mean office systolic BP levels (in mm Hg) in the sitting position among the patients with HT and CAD recieved the biso/perindopril FDC
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
mm Hg
  SBP | -24.92 (16.43)
  DBP | -12.21 (11.03)

2. Secondary Outcome: Change in Mean Systolic and Diastolic BP Levels at Week 4 Compared With Baseline.
Description: Change in mean systolic and diastolic BP levels at week 4 of treatment with SPC compared with baseline.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
mm Hg
  Systolic BP | -17.32 (13.97)
  Dyastolic BP | -8.39 (8.79)

3. Secondary Outcome: Change in Number of Angina Attacks Per Week at Week 4 Compared With Baseline.
Description: Change in number of angina attacks per week at week 4 of treatment compared with baseline.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: angina attacks per week
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
angina attacks per week | 2.76 (2.26)

4. Secondary Outcome: Change in Number of Angina Attacks Per Week at Week 12 Compared With Baseline
Description: Change in number of angina attacks per week at week 12 of treatment compared with baseline.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: angina attacks per week
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
angina attacks per week | 0.95 (0.94)

5. Secondary Outcome: Proportion of Patients Who Were Taking Lipid Lowering Therapy
Description: Proportion of patients who were taking lipid lowering therapy (LLT) at week 12 of treatment
Time Frame: 3 months
Measure: Number; unit: Number of Participants Who Were Taking L
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 463
Number of Participants Who Were Taking L | 397

6. Secondary Outcome: SBP ≤140 mm Hg and DBP ≤90 mm Hg at Week 4 Compared With Baseline
Description: Proportion of patients who achieved SBP ≤140 mm Hg and DBP ≤90 mm Hg at week 4.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
Participants | 330

7. Secondary Outcome: SBP ≤140 mm Hg and DBP ≤90 mm Hg at Week 12 Compared With Baseline
Description: Proportion of patients who achieved SBP ≤140 mm Hg and DBP ≤90 mm Hg at week 12
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
Participants | 417

8. Secondary Outcome: Younger Than 65 Who Achieved SBP ≤130 mm Hg and DBP ≤80 mm Hg at Week 4 of Treatment Compared With Baseline
Description: Proportion of patients younger than 65 who achieved SBP ≤130 mm Hg and DBP ≤80 mm Hg at week 4 of treatment
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 295
Participants | 86

9. Secondary Outcome: Younger Than 65 Who Achieved SBP ≤130 mm Hg and DBP ≤80 mm Hg at Week 12 of Treatment
Description: Proportion of patients younger than 65 who achieved SBP ≤130 mm Hg and DBP ≤80 mm Hg at week 12 of treatment.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 293
Participants | 143

10. Secondary Outcome: Older Than 65 Years Who Achieved SBP≤140 mm Hg and DBP ≤90 mm Hg at Week 4 of Treatment
Description: Proportion of patients older than 65 years who achieved SBP≤140 mm Hg and DBP ≤90 mm Hg at week 4 of treatment
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 186
Participants | 109

11. Secondary Outcome: Older Than 65 Years Who Achieved SBP≤140 mm Hg and DBP ≤90 mm Hg at Week 12 of Treatment
Description: Proportion of patients older than 65 years who achieved SBP≤140 mm Hg and DBP ≤90 mm Hg at week 12 of treatment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 186
Participants | 162

12. Secondary Outcome: Mean Heart Rate (HR) at Week 4 Compared With Baseline.
Description: Changes in the mean heart rate (HR) at week 4 of treatment compared with baseline
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
beats per minute | -10.87 (10.36)

13. Secondary Outcome: Mean Heart Rate (HR) at Week 12 Compared With Baseline.
Description: Changes in the mean heart rate (HR) at week 12 of treatment compared with baseline
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
beats per minute | -14.44 (11.69)

14. Secondary Outcome: Patients Who Achieved Target Level of Resting HR (55-60 Bpm) at Week 4
Description: Proportion of patients who achieved target level of resting HR (55-60 bpm) at week 4 of treatment.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
Participants | 82

15. Secondary Outcome: Patients Who Achieved Target Level of Resting HR (55-60 Bpm) at Week 12
Description: Proportion of patients who achieved target level of resting HR (55-60 bpm) at week 12 of treatment.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAD Patients With Previous MI and HTN
Number analyzed (Participants) | 481
Participants | 150

ADVERSE EVENTS:
Time Frame: 3 month
Arm/Group | CAD Patients With Previous MI and HTN
All-Cause Mortality (participants affected / at risk) | 0/504
Serious Adverse Events (participants affected / at risk) | 0/504
Other Adverse Events (participants affected / at risk) | 0/504

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04656847/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04656847/ICF_001.pdf